CLINICAL TRIAL: NCT06692686
Title: The Development of Patient-Centered Clinical AFO Prescription Guidelines to Optimize Post-Stroke Function and Quality of Life
Brief Title: AFO Prescription to Optimize Post-Stroke Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Medical University of South Carolina (Other); Rancho Los Amigos National Rehabilitation Center (Other); Hanger Clinic: Prosthetics & Orthotics (Other); Brooks Rehabilitation (Other)
Responsible Party: Principal Investigator, Rick Neptune, Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006128; CDMRP-OP230030 (Other Grant/Funding Number: DoD - USAMRAA)
Record Dates: First submitted 2024-11-07; First posted 2024-11-18 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ankle Foot Orthosis (AFO); Stroke Patients; Post-Stroke Hemiparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- PF-CS-MA (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the pre-fabricated (PF) AFO, followed by the carbon strut (CS) AFO, and finally the multifunctional articulating (MA) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)
- PF-MA-CS (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the pre-fabricated (PF) AFO, followed by the multifunctional articulating (MA) AFO, and finally the carbon strut (CS) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)
- CS-PF-MA (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the carbon strut (CS) AFO, followed by the pre-fabricated (PF) AFO, and finally the multifunctional articulating (MA) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)
- CS-MA-PF (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the carbon strut (CS) AFO, followed by the multifunctional articulating (MA) AFO, and finally the pre-fabricated (PF) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)
- MA-PF-CS (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the multifunctional articulating (MA) AFO, followed by the pre-fabricated (PF) AFO, and finally the carbon strut (CS) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)
- MA-CS-PF (Experimental): Participants will wear each of the three ankle-foot orthosis (AFO) treatment options over three separate four-week periods. In this arm, participants first use the multifunctional articulating (MA) AFO, followed by the carbon strut (CS) AFO, and finally the pre-fabricated (PF) AFO.
  Interventions: Device: Pre-fabricated (PF) ankle-foot orthosis (AFO); Device: Carbon-strut (CS) ankle-foot orthosis (AFO); Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO)

INTERVENTIONS:
Device: Pre-fabricated (PF) ankle-foot orthosis (AFO) — These pre-manufactured orthoses are customized to fit each patient. These devices can help to distribute weight evenly along the foot, but do not offer much opportunity for adjustment to a patient's specific needs. These AFOs achieve ankle motion through material deflection and lack a single point of articulation.
Device: Carbon-strut (CS) ankle-foot orthosis (AFO) — These AFO designs are built from a custom mold of the patient's affected limb for a more individualized fit. It includes a solid ankle design and achieves ankle motion through material deflection and lacks a single point of articulation.
Device: Multifunctional articulating (MA) ankle-foot orthosis (AFO) — These AFO designs are also built from a custom mold of the patient's affected limb, but these orthoses have a true articulation at the ankle to provide controlled ankle movement in a range determined appropriate by the orthotist through gait analysis.

SUMMARY:
The overall goal of this study is to attain the highest possible health-related quality of life for individuals with lower-limb impairment through a clinical trial examining three different modern carbon fiber ankle-foot orthosis (AFO) treatment options targeting the rehabilitation of individuals post-stroke. To achieve this goal, the investigators will:

1. Identify the factors that significantly contribute to an individual's highest potential quality of life when considering each of the three available AFO design options, and
2. Develop prediction models of clinical performance using biomechanical function linked to the three AFO designs.

Participants will be asked to:

* Wear each of the three modern AFO designs for one month, after receiving therapy training and
* Complete questionnaires and performance tests with each AFO.

In addition, the subset of individuals participating in goal 2) will also be asked to:

* Perform biomechanical analyses using high-speed cameras and force plates during different walking and balance tests with each AFO design.

ELIGIBILITY:
Inclusion Criteria:

* be a minimum of three months post-stroke
* be greater than 18 years of age
* have been prescribed either a semi-rigid or a custom-made articulating AFO
* wear their prescribed AFO for all primary mobility activity outside the house
* be able to walk at least 20 meters without manual assistance
* walk at least 10 meters per minute (12% of normal velocity) during a 6-meter self-selected velocity walking test.

Exclusion Criteria:

* having a condition that could significantly limit ambulation, including severe osteoarthritis, rheumatoid arthritis, congestive heart failure, or pre-existing neurological disorder other than post-stroke
* having cognitive deficits that preclude their ability to provide consent for participation
* having an ankle plantar flexion contracture equal to or greater than 15 degrees plantar flexion with full knee extension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | Over the real-world use period (4 weeks) for each AFO
  Health-related quality of life (HRQoL) is a framework that considers physical, mental, emotional, and social function when assessing the satisfaction of AFO users with their AFO.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rancho Research Institute, Downey, California
  - Brooks Rehabilitation, Jacksonville, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - Hanger Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Final research de-identified data generated from this project will be made available to the research community upon request. Data requests may be subject to a signed data user agreement (DUA).

REFERENCES:
- [Background] Wilson IB, Cleary PD. Linking clinical variables with health-related quality of life. A conceptual model of patient outcomes. JAMA. 1995 Jan 4;273(1):59-65. PMID 7996652